CLINICAL TRIAL: NCT03407443
Title: Evaluation of the VA's Public Awareness Campaigns
Brief Title: Pilot the Use of VA Make the Connection Campaign to Facilitate Help Seeking Among Vulnerable Veterans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Canandaigua VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Karras, Health Science Specialist, Canandaigua VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB899190
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mental Health Issue (E.G., Depression, Psychosis, Personality Disorder, Substance Abuse); Help-Seeking Behavior
Keywords: mental health promotion campaign; veterans
MeSH Terms: conditions — Depression; Psychotic Disorders; Personality Disorders; Substance-Related Disorders; Help-Seeking Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exposure to Make the Connection messages (Experimental)
  Interventions: Other: Exposure to Make the Connection messages
- Active Control group (Active Comparator)
  Interventions: Other: Active Control Group
- No exposure control group (No Intervention)

INTERVENTIONS:
Other: Exposure to Make the Connection messages — Participants are exposed to Make the Connection messages (each approximately 3 minutes in length) weekly for over a four-month study period through the study mobile application.
  Arms: Exposure to Make the Connection messages
Other: Active Control Group — Participants are exposed to VA news clips/segments (each approximately 3 minutes in length) weekly for over a four-month study period through the study mobile application.
  Arms: Active Control group

SUMMARY:
This pilot study seeks to determine if exposure to the Make the Connection campaign messages developed by the U.S. Department of Veterans Affairs (VA) is associated with changes in mental-health related outcomes, specifically: (1) psychosocial determinants that drive help seeking behaviors (knowledge, attitudes and intentions); and (2) perceived barriers to seeking care. Participants are randomly assigned to message exposure or control (no exposure) conditions. Data from this project will inform mental health education and outreach efforts targeted towards Veterans experiencing mental health concerns.

ELIGIBILITY:
Inclusion Criteria:

Veterans of all gender/sex, race/ethnicities that in the past 6 months:

* utilized health services in the U.S. Department of Veterans Affairs (VA);
* screened positive on the PHQ-2, AUDIT-C or PC-PTSD and/or received a mental health diagnosis as documented in VA medical record
* Fluent in English language
* Capable of understanding goals of study
* Capable of providing verbal consent
* Willing and able to download/use study Android mobile application for duration of study

Exclusion Criteria:

* Not a U.S. Veteran who has utilized VA health care in the past 6 months
* Did not screen positive and/or was not diagnosed with mental health disorder
* Determined cognitively impaired and unable to provide verbal consent
* Determined to be in high distress during recruitment screening
* Currently institutionalized (i.e., hospitalized; incarcerated, etc.)
* Unwilling and/or unable to download and use use the study app

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
change in help seeking behavior | change from baseline behavior at 16 weeks
  self-report treatment engagement in VA or non-VA services

SECONDARY OUTCOMES:
Attitudes towards help seeking | assessed up to 16 weeks
  self-reported treatment beliefs and likelihood for help seeking
Barriers to care | assessed up to 16 weeks
  The 6-item stigma Scale developed by Britt et al. (2000; 2008) to assess stigma of accessing treatment for psychological problems among military personnel is used w/a 5 point likert scale (1=strongly disagree to 5=strongly agree). Logistical barriers to care are also assessed using the 5-item Barriers to Care scale (Hoge et al. 2004) to assess barriers to accessing psychological treatment w/ a 5 point likert scale (1=strongly disagree; 5= strongly agree). Higher values represent a worse outcome (e.g., higher endorsement of stigma).

OTHER OUTCOMES:
change in social support | change from baseline behavior at 16 weeks
  self-report survey using the multidimensional scale of perceived social support (Zimmet et al. 1990). This is a 12-item scale of perceived social support from family and friends. Each item is scored 1-7 on a likert scale (1=very strongly disagree; 7=very strongly agree) and summed with a possible range of 7 to 84. Higher scores indicate higher awareness/belief of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Karras, PhD, Principal Investigator — Center of Excellence for Suicide Prevention, Canandaigua VA Medical Center; U.S. Department of Veterans Affairs